CLINICAL TRIAL: NCT06437093
Title: The Effect of Relactation Support Program on Milk Release, Mother-Infant Attachment and Maternity Role
Brief Title: The Effect of Relactation Support Program on Milk Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Emel GÜÇLÜ CİHAN, Principal Investigator, Inonu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: emelabdullahyusuf46
Record Dates: First submitted 2024-01-09; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Breast Feeding, Exclusive; Mother-Child Relations
Keywords: breast feeding; connecting; maternal role
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: This is a single-group pre-test post-test experimental study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-group pre-test post-test experimental study (Experimental): In our midwifery intervention, the mother was firstly educated about breastfeeding and relactation, using educational brochures prepared by the researchers. Afterwards, the mother was taught "nipple stimulation", "skin-to-skin contact" and "finger feeding method", and the first feeding of the baby was performed together with the mother. After this first intervention in the FHC, all interventions were performed at home. The follow-ups continued for 15 days with one day of telephone support and one day of home visit. Since the majority of mothers did not accept video calls (privacy, etc.), telephone support was provided only verbally.
  Interventions: Other: TEACHING RELACTATION TECHNIQUES

INTERVENTIONS:
Other: TEACHING RELACTATION TECHNIQUES — In our midwifery intervention, the mother was firstly educated about breastfeeding and relactation, using educational brochures prepared by the researchers. Afterwards, the mother was taught "nipple stimulation", "skin-to-skin contact" and "finger feeding method", and the first feeding of the baby was performed together with the mother. After this first intervention in the FHC, all interventions were performed at home. The follow-ups continued for 15 days with one day of telephone support and one day of home visit. Since the majority of mothers did not accept video calls (privacy, etc.), telephone support was provided only verbally.
  Other Names: BREASTFEEDING EDUCATION

SUMMARY:
Aim: This study aimed to determine the effect of relactation support program on milk release, mother-infant attachment and maternity role.

Materials and Methods: This single-group pre-test post-test experimental study was conducted with 34 mothers who had 1-4 month old infants, stopped breastfeeding at least 15 days and at most 3 months ago and were registered in the family health centers of a province in the southern Turkey. The relactation support program was completed in 15 days, with eight home visits and seven telephone support sessions. The data were collected using a personal information form, a mother-infant follow-up form, the Maternal Attachment Inventory (MAI) and the Barkin Index of Maternal Functioning (BIMF).

Keywords: Mother-Infant Attachment, Maternity Role, Midwifery, Relactation, Milk Release.

DETAILED DESCRIPTION:
This is a single-group pre-test post-test experimental study. This study was conducted between October 2021 and October 2022 in Family Health Centers (FHCs) in province in southern Turkey. By using the G*power 3.1 program, the sample size was determined to include 29 mothers/women under 5% margin of error, 95% confidence level, and 95% power of representation.

ELIGIBILITY:
Inclusion Criteria:

For mothers;

* Having no milk release,
* Using no pharmacological agents that may increase milk release,
* Being not pregnant,
* Having no communication problem,
* Being literate,
* Being between the ages of 18-35 years,
* Having singleton gestation in their last childbirth,
* Using no medication that prevents breastfeeding (chemotherapy, etc.). For babies;
* Being healthy
* Having no congenital sucking problem (cleft palate, cleft lip, etc.)

Exclusion Criteria:

For mothers;

* Using any pharmacologic agent to increase milk release,
* Having a diagnosis of psychiatric illness. For babies;
* Having any metabolic disease that may prevent breastfeeding (galactosemia, phenylketonuria, etc.) or any other chronic disease (advanced heart disease, etc.).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Questionnaire | First day
  Mother-Infant Follow-Up Form filled out at the first meeting with the participants.This form was prepared by the researchers and includes information about the mothers' breastfeeding issues, breast health problems (cracks, mastitis, etc.), number of daily breastfeeding, number of daily milk release, amount of milk release, baby's weight and presence of sucking problems, which should be followed up during relactation.
Scale 1 | First day
  Maternal Attachment Scale was used for pretest.This 4-point Likert-type scale has a total of 26 items, scoring as "always =4", "often =3", "sometimes =2", and "never =1". The lowest and highest scores on the scale are 26 and 104, respectively. Higher scale scores refer to greater maternal attachment.
Scale 2 | First day
  Barkin Index of Maternal Functioning Scale was used for pretest. Index of Maternal Functioning consists of 16 items, scoring as "completely disagree=0", "disagree=1", "partially disagree=2", "undecided=3", "partially agree=4", "agree=5", "completely agree=6". The lowest and highest scores on the scale are 0 and 96, respectively. The scale has five subscales:
  * Self-Care (2, 11, 13 items)
  * Maternal Psychology (8, 10 items)
  * Infant Care (items 12, 14, 15, 16)
  * Social Support (items 6, 7, 9)
  * Maternal adjustment (items 1, 3, 4, 5).

SECONDARY OUTCOMES:
Questionnaire | 1-16 days
  Mother-Infant Follow-Up Form was filled out every day for 15 days.Finally, it was filled on the 16th day.
Scale 1 Scale 1 (Attachment Inventory) | 16. day
  Maternal Attachment Scale was used for posttest.
Scale 2 | 16. day
  The Barkin Index of Maternal Functioning was used for posttest.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu Universty, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No